CLINICAL TRIAL: NCT01873846
Title: A Study to Evaluate the Product Performance of a New Silicone Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 817
Record Dates: First submitted 2013-05-28; First posted 2013-06-10 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Silicone Hydrogel Contact Lens (Experimental): Contact lenses to be worn in each eye on a daily wear basis for 2 weeks. Participants will be provided with Bausch + Lomb Biotrue® multi-purpose solution and contact lens cases for daily rinsing, cleaning, disinfecting, and storing their lenses.
  Interventions: Device: Silicone Hydrogel Contact Lens

INTERVENTIONS:
Device: Silicone Hydrogel Contact Lens

SUMMARY:
The objective of this study is to evaluate the product performance of a new silicone hydrogel soft contact lens when worn by current soft contact lens wearers on a daily wear basis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be correctable through spherocylindrical refraction to 32 letters (0.3 logMAR) or better (distance, high contrast) in each eye
* Subjects must have clear central corneas and be free of any anterior segment disorders.
* Subjects must be adapted lens wearers and wear a lens in each eye and each lens must be of the same manufacture and brand.
* Subjects must be myopic and require lens correction from -0.25 D to -6.00 D in each eye.
* Subject must wear their current lenses for a minimum of 12 hours per day at least four days per week.
* Subjects must spend at least 3 hours each workday using a computer or electronic device (ie, smartphones, tablets, eReaders).
* Subjects must habitually wear soft contact lens.
* Subject must have no active ocular disease or allergic conjunctivitis.
* Subject must not be using any topical ocular medications.
* Subjects must be bothered (occasionally or frequently) by blurriness or fluctuations in vision with their current contact lenses.
* Subjects must habitually use a lens care product for cleaning, disinfection, and storage.

Exclusion Criteria:

* Subjects who have worn gas permeable (GP) contact lenses within the last 30 days or who have worn polymethylmethacrylate (PMMA) lenses within the last three months.
* Subjects with any systemic disease currently affecting ocular health or which in the Investigator's opinion may have an effect on ocular health during the course of the study.
* Subjects using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Subjects with an active ocular disease or who are using any ocular medication.
* Subjects who are not correctable to 32 letters (0.3 logMAR) in each eye with soft spherical contact lenses.
* Subjects who are presbyopic or currently wear monovision, multifocal, or toric contact lenses.
* Subjects with an ocular astigmatism of 1.00 D or greater in either eye.
* Subjects with anisometropia (spherical equivalent) of 2.00 D or greater in either eye.
* Subjects with any Grade 2 or greater finding during the slit lamp examination.
* Subjects with corneal infiltrates, of ANY GRADE, are not eligible.
* Subjects with any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Subjects with any scar or neovascularization within the central 4 mm of the cornea.
* Subjects who are aphakic.
* Subjects who are amblyopic.
* Subjects who have had any corneal surgery (eg, refractive surgery).
* Subjects who are allergic to any component in the study care products.
* Subjects who are bothered by blurriness or fluctuations in vision due to itchy eyes, something on or under the lens, allergies, or cigarette smoke.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Varughese, Study Director — Valeant Pharmaceuticals
Locations (1):
- Bausch & Lomb Incorporated, Madison, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Silicone Hydrogel Contact Lens: Contact lenses to be worn in each eye on a daily wear basis for 2 weeks. Participants will be provided with Bausch + Lomb Biotrue® multi-purpose solution and contact lens cases for daily rinsing, cleaning, disinfecting, and storing their lenses.
  Silicone Hydrogel Contact Lens
Period: Overall Study
Arm/Group | Silicone Hydrogel Contact Lens
Started | 400
Eligble Participants Dispensed Lenses | 396
Completed | 388
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: Eligible participants dispensed lenses
Arm/Group | Silicone Hydrogel Contact Lens
Number analyzed (Participants) | 396
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 278
  Male | 118
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 44
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 14
  White | 327
  More than one race | 0
  Unknown or Not Reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Preference Question: How Would You Say These Contact Lenses Compare Overall With the Contact Lenses You Usually Use?
Description: Participants will respond to a survey regarding their experience wearing the Test Lens after 7 days of wear. Participants were asked to answer the following question: "How would you say these contact lenses compare overall with the contact lenses you usually use?" Prefer study lenses Prefer usual lenses About the same as usual lenses
Time Frame: 7 days
Population: There were 380 eligible subjects with lenses dispensed.
Measure: Count of Participants; unit: Participants
Arm/Group | Silicone Hydrogel Contact Lens
Number analyzed (Participants) | 380
Participants
  Prefer study lenses | 195
  Prefer usual lenses | 93
  About the same as usual lens | 92

2. Primary Outcome: Preference Question: These Contact Lenses Deliver Exceptional Clarity and Comfort All Day Long.
Description: Participants will respond to a survey regarding their experience wearing the Test Lens after 7 days of wear. Participants were asked to assess the following statement with respect to their usual contact lenses: "These contact lenses deliver exceptional clarity and comfort all day long." Prefer study lenses Prefer usual lenses About the same as usual lenses
Time Frame: 7 days
Population: There were 380 eligible subjects with lenses dispensed.
Measure: Count of Participants; unit: Participants
Arm/Group | Silicone Hydrogel Contact Lens
Number analyzed (Participants) | 380
Participants
  Prefer study lenses | 199
  Prefer usual lenses | 80
  About the same as usual lens | 101

3. Primary Outcome: Preference Question: These Contact Lenses Help Maintain Healthy, White Eyes.
Description: Participants will respond to a survey regarding their experience wearing the Test Lens after 7 days of wear. Participants were asked to assess the following statement with respect to their usual contact lenses: "These contact lenses help maintain healthy, white eyes." Prefer study lenses Prefer usual lenses About the same as usual lenses
Time Frame: 7 days
Population: There were 380 eligible subjects with lenses dispensed.
Measure: Count of Participants; unit: Participants
Arm/Group | Silicone Hydrogel Contact Lens
Number analyzed (Participants) | 380
Participants
  Prefer study lenses | 162
  Prefer usual lenses | 51
  About the same as usual lens | 167

4. Secondary Outcome: Lens Performance Assessment
Description: High Contrast Distance logMAR Lens VA Change From Baseline to Week 2.
Time Frame: 2 weeks
Population: High contrast distance lens visual acuity (VA) was assessed at Screening/Dispensing on the Test (newly dispensed) lenses, and at the follow-up visit(s). The population included subjects with baseline and at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Log of Minimum Angle of Resolution VA
Units Other Than Participants: Eyes
Arm/Group | Silicone Hydrogel Contact Lens
Number analyzed (Participants) | 382
Number analyzed (Eyes) | 764
Log of Minimum Angle of Resolution VA | 0.004 (0.067)

5. Secondary Outcome: Any Graded Slit Lamp Finding > 2
Description: Slit lamp findings for each eye, including epithelial edema, epithelial microcysts, corneal staining, limbal and bulbar injections, upper lid tarsal conjunctival abnormalities, corneal neovascularization, and corneal infiltrates, were graded for severity on a scale from 0 (No Finding) to 4 (Severe Finding). Corneal staining grades were computed as the maximum grade over grades taken within each of five different eye locations (central, inferior, nasal, superior, and temporal). Eyes with multiple visits are counted once for the highest grade.
Time Frame: 2 weeks
Population: Percentages are based on the number of dispensed eyes with non-missing scores.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Silicone Hydrogel Contact Lens
Number analyzed (Participants) | 396
Number analyzed (Eyes) | 792
Eyes | 2

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Silicone Hydrogel Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/396
Other Adverse Events (participants affected / at risk) | 0/396

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No